CLINICAL TRIAL: NCT00224783
Title: Placebo-controlled Double-blind Controlled Trial of Single Intranasal Inoculation of CAIV-T Liquid Formulation in Healthy Japanese Male Adults
Brief Title: Phase I Trial Evaluating Safety and Tolerability of CAIV-T in Healthy Japanese Male Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Christopher Ambrose, MD, Medimmune, LLC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D153 P800; NCT00192530 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-23 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Japanese Male Adults
MeSH Terms: interventions — FluMist

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAIV-T (Active Comparator): CAIV-T contains 3 cold-adapted influenza virus strains (A/H1N1, A/H3N2, B) concentrated and refined by centrifugal separation from the chorioallantoic membrane of specific pathogen-free (SPF) eggs, containing SPG (sucrose-phosphate-glutamate), arginine, and acid hydrolyzed pig gelatin as stabilizers. Subjects were inoculated once with about 0.1 mL of investigational vaccine in each nasal cavity (a total of 0.2 mL) using a nebulizer.
  Interventions: Biological: CAIV-T
- Placebo (Placebo Comparator): Placebo contained 0.01 mol/L potassium phosphate buffer containing 0.85% sodium chloride (pH 7.2). Subjects received about 0.1 mL (a total 0.2 mL) of the control drug using a nebulizer.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CAIV-T — Trivalent cold adapted temperature sensitive attenuated Types A and Type B influenza virus live vaccine (CAIV-T)
  Other Names: 0.2 mL, by nebulizer
  Arms: CAIV-T
Biological: Placebo — 0.2 mL of 0.01 mol/L potassium phosphate buffer containing 0.85% sodium chloride (pH 7.2).
  Arms: Placebo

SUMMARY:
The primary objective of the study was to investigate the safety and tolerability of CAIV-T liquid formulation in healthy Japanese male adults.

DETAILED DESCRIPTION:
The primary objective of the study was to investigate the safety and tolerability of CAIV-T liquid formulation in healthy Japanese male adults by evaluating the incidence of influenza-like symptoms, and the type, incidence, and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 years old or over but below 45 years old (at the time of consent)
* Persons judged suitable by the principal investigator or investigator from the results of prior history, physical examination and clinical findings.
* Persons having the ability to understand consent and a written consent obtained prior to the start of screening.
* Persons being able to participate in the trial for 1 month from the inoculation of the trial vaccine to the completion of the trial.
* Persons being able to be contacted (by phone, hospital visit or house visit) by the trial staff at the time of testing after 28 days from the inoculation of the trial vaccine.

Exclusion Criteria:

* Persons judged to be impossible or difficult to contact for requesting hospital visits to carry out clinical evaluation and tests during the trial term.
* Persons having a prior history of or suspected immunological disease, or those receiving administration of systemic corticosteroids or immunosuppressants such as cytotoxic drugs (e.g., methotrexate, etc.)
* Persons having blood formulations such as immunoglobulin, etc., administered or planned during a period from one month before the inoculation of the trial vaccine to the completion of the trial.
* Persons living with any person with a nonfunctional or suppressed immune system (by using immunosuppressants, etc.), in the same household.
* Persons with a prior history of hypersensitivity to chicken eggs or chicken egg proteins or components of the trial vaccine (such as sucrose, phosphoric acid, glutamate, arginine and acid-hydrolyzed pig gelatin).
* Persons inoculated with a live virus vaccine within 1 month before screening.
* Persons having the planned administration of another trial vaccine or drug during the period from one month before screening to the completion of the trial
* Person having an influenza treatment drug (such as commercially available drugs or trial vaccines: for example, Oseltamivir, Zanamivir, Amantadine, etc.), administered within one month before screening. Incidentally, no prophylactic administration of an influenza viral drug was permitted.
* Persons inoculated with an influenza vaccine within 6 months before screening or planned to be inoculated with an influenza vaccine during the term of the present trial.
* Persons with blood drawn quantity (including blood donation) of 400 mL or more within 3 months or 200 mL or more within 1 month before screening.
* Persons with a history of any febrile disorders (oral cavity temperature ³ 38.0°C) or other acute disorders within 36 hours before trial vaccine inoculation.
* Persons who had upper respiratory tract disorders themselves or whose family members had such disorders within 72 hours before trial vaccine inoculation.
* Persons treated with an antibiotic within 72 hours before trial vaccine inoculation.
* Persons with an acute asthmatic symptom.
* Persons judged to have a pathology preventing the evaluation of the trial effect by the principal investigator (or investigator).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2002-08; Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
The number of subjects within each treatment arm who experienced influenza-like symptoms | Within 6 days post vaccination
  Influenza-like symptoms, ie, typical clinical symptoms of influenza infection, including fever (oral temperature > or = 38 degrees C), cough, runny or stuffy nose, sore throat, headache, chills, muscular pain, vomiting, decline in activity, decline in appetite.

SECONDARY OUTCOMES:
The number of subjects within each treatment arm who experienced adverse events | Within 28 days of vaccination
  Adverse events were classified according to the "Glossary of Side Effects of Pharmaceutical Agents, 1996."

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC